CLINICAL TRIAL: NCT06995339
Title: Comparative Clinical and Biochemical Study Evaluating the Effectiveness of Metformin Versus Febuxostate on Gouty Obese Non-Diabetic Patients
Brief Title: Comparative Clinical and Biochemical Study Evaluating the Effectiveness of Metformin Versus Febuxostat on Gouty Obese Non-Diabetic Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Dalia Naser Abdel-Sadek Safa , Faculty of Pharmacy, Tanta University (Unknown); Sahar Mohamed Elhaggar, Faculty of Pharmacy, Tanta University (Unknown); Tarek Mohamed Abd-Elazez Nasr-Allah, Faculty of Medicine - Al-Azhar University (Unknown)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58479
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Febuxostat; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): patients will receive febuxostat 80 mg daily for 6 months.
  Interventions: Drug: Febuxostat Tablets
- Metformin group (Active Comparator): patients will receive metformin 1000 mg daily for 6 months
  Interventions: Drug: Febuxostat Tablets; Drug: Metformin

INTERVENTIONS:
Drug: Febuxostat Tablets — Febuxostat is a selective xanthine oxidase inhibitor (XOI) that targets uric acid generation. It has been used as a SUA lowering agent in patients not responding to allopurinol
Drug: Metformin — Metformin is an oral antihyperglycemic drug widely used in type 2 diabetes (T2DM) treatment. Most of its effects are exerted via an indirect induction of the phosphorylated activation of AMP-activated protein kinase (AMPK)
  Arms: Metformin group

SUMMARY:
Gout is a systemic disease that results from the deposition of monosodium urate crystals (MSU) in tissues. Increased serum uric acid (SUA) above a specific threshold (>6.8 mg/dl) is a requirement for the formation of uric acid crystals. MSU crystals can be deposited in all tissues mainly in and around the joints forming tophi. Early presentation of gout is an acute joint inflammation that is quickly relieved by non-steroidal anti-inflammatory drugs (NSAIDs) or colchicine. Lowering SUA levels below deposition threshold either by dietary modification or using serum uric acid lowering drugs is the main goal in management of gout. This results in dissolution of MSU crystals preventing further attacks

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged < 18 years.
* All patients are diagnosed to have gout with serum uric acid < 7 mg/dl.
* All patients are diagnosed to have obesity with body mass index (BMI) ≥ 30 kg/m2.

Exclusion Criteria:

* The presence of any type of diabetes mellitus.
* Patients with drug-induced hyperuriceamia (those taking anti-TB agents, low dose aspirin, cytotoxic chemotherapy, diuretics, immunosuppressants, fructose, lactate infusion, testosterone or xylitol).
* Non-obese patients with BMI >30 kg/m2.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in serum uric acid level | 3 months
  Serum uric acid is the major metabolite of purine pathway and used in diagnosis of gouty patients

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt